CLINICAL TRIAL: NCT03724617
Title: Clinical Study of Stem Cells in the Treatment of Thin Endometrium
Brief Title: Clinical Study of Umbilical Cord Mesenchymal Stem Cells Combined With Collagen Scaffold in the Treatment of Thin Endometrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xiaona Lin, senior doctor, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRSHRMC20180924
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2018-10

CONDITIONS: Thin Endometrium; Intrauterine Adhesion
Keywords: thin endometrium; Intrauterine Adhesion; stem cell; Collagen scaffold
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stem cell therapy (Experimental)
  Interventions: Drug: umbilical cord mesenchymal stem cells combined with collagen scaffold

INTERVENTIONS:
Drug: umbilical cord mesenchymal stem cells combined with collagen scaffold — 3-7 days after the end of menstruation, we underwent hysteroscopic exploration and separation if there was intrauterine adhesions. Intraoperative endometrial biopsy, recording biopsy location, endometrial specimens sent to HE examination and immunohistochemistry (vwf detection of microvessel density). The umbilical cord mesenchymal stem cell combined with collagen scaffold was spread on the balloon scaffold and placed in the uterine cavity. 5 ml of saline was filled into the balloon, and B-ultrasound confirmed that the scaffold was attached to the uterine wall. The patient was hospitalized for 2 hours and the patient's vital signs were recorded.

SUMMARY:
This is a non-blind self-control trial. We mainly compare the changes of endometrial thickness，changes in menstrual flow, and improvement in pregnancy before and after stem cell treatment in patients with thin endometrium.

DETAILED DESCRIPTION:
According to the medical history and the results of the examination, the selected cases were screened and the informed consent was signed. After hysteroscopy, the collagen/umbilical cord mesenchymal stem cell was spread on a foley catheter, and placed in the uterine cavity, and 5 ml of saline was filled into the balloon. B-ultrasound confirmed that the stent was attached to the uterine wall. The balloon was removed in situ after 1 week. We mainly compare the endometrial thickness before and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. According to the GCP regulations, obtain the informed consent of the subject, volunteer for the test, and have signed the informed consent form.
2. Women aged 20-40 years with fertility requirements
3. Infertility patients who are treated in this hospital
4. After more than 2 times of hysteroscopic adhesion separation surgery, the uterine cavity morphology has basically returned to normal. The patient has a normal menstrual cycle or an estrogenic dose of 6 mg per day, and the highest thickness of the endometrium is 5.5 mm in 6 cycles by ultrasound.
5. or receive adjuvant reproductive treatment, the endometrial thickness is less than 5.5mm for unknown reasons, the treatment of estrogen, colony stimulating factor, aspirin, sildenafil and other drugs up to 8mg / day is invalid.
6. HBVAg negative, HCV negative, HIV negative, syphilis negative
7. Normal bone marrow morphology, normal blood routine
8. Previously failed to receive relevant stem cell therapy

Exclusion Criteria:

1. Those who cannot accept the treatment observation process required by the test
2. There are contraindications for hysteroscopic surgery;
3. congenital uterine malformation; severe adenomyosis; uterine fibroids that may affect embryo implantation; the investigators judged that there are other uterine factors that are not suitable for embryo implantation
4. Patients with chromosomal abnormalities
5. contraindications to estrogen therapy; systemic diseases such as thrombosis, cardiopulmonary disease, hematopoietic diseases, malignant tumors, etc.
6. Patients without fertility requirements

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
the change of endometrial thickness | Change from Baseline endometrial thickness at 6 months
  B-ultrasound measures and compares the endometrial thickness of the luteal phase before and after administration.

SECONDARY OUTCOMES:
pregnancy rate | pregnancy rate at 1 year
  pregnancy rate = (pregnancy / observations) × 100%
live birth rate | live birth rate at 1 year
  live birth rate = (live births / observations) × 100%
abortion rate | abortion rate at 1 year
  abortion rate = (number of abortions / observations) × 100%

CONTACTS AND LOCATIONS:
Overall Officials: Xiaona Lin, Study Chair — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw hopital,School of medicine,Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Shi L, Lin X, Zhou F, Xin L, Xu W, Yu H, Li J, Pan M, Pan Y, Dai Y, Zhang Y, Shen J, Zhao L, Lu M, Zhang S. Unresponsive thin endometrium caused by Asherman syndrome treated with umbilical cord mesenchymal stem cells on collagen scaffolds: a pilot study. Stem Cell Res Ther. 2021 Jul 22;12(1):420. doi: 10.1186/s13287-021-02499-z. PMID 34294152